CLINICAL TRIAL: NCT02690779
Title: Impact of a Patient Educational Video on Bowel Preparation Quality for Screening Colonoscopy: a Quality Assurance Project
Brief Title: Bowel Preparation Quality for Screening Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Keith Obstein, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 131668
Record Dates: First submitted 2016-01-19; First posted 2016-02-24 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Screening Colonoscopies
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients watching educational video (Experimental): The educational intervention will consist of a 2-3 minute video demonstrating video images of adequate and inadequate bowel preps, and reviewing instructions for split dose prep administration. This video will be posted on YouTube. Group 1 will consist of 30 subjects who will be instructed to view this video prior to beginning their colonoscopy preparation. Information to access the YouTube video will be provided to the patients by endoscopy nurse assessment staff when contacting the patients as per standard practice to review appointment scheduling and procedure-day logistics.
  Interventions: Other: Educational intervention
- Patients not watching educational video (Sham Comparator): Group 2 will consist of 30 subjects who will not receive instructions to view the video. They will be given routine care instructions for bowel prep.
  Interventions: Other: Routine Care Instructions

INTERVENTIONS:
Other: Educational intervention — 2-3 minute video demonstrating video images of adequate and inadequate bowel preps, and reviewing instructions for split dose prep administration.
  Arms: Patients watching educational video
Other: Routine Care Instructions — patients will follow routine care and instructions
  Arms: Patients not watching educational video

SUMMARY:
The study will consist of a prospective observational period performed in the GI Endoscopy Lab. The objective is to document the quality of bowel preps in patients undergoing a screening colonoscopy with and without an educational intervention.

DETAILED DESCRIPTION:
The educational intervention will consist of a 2-3 minute video demonstrating video images of adequate and inadequate bowel preps, and reviewing instructions for split dose prep administration. This video will be posted on YouTube. Group 1 will consist of 30 subjects who will be instructed to view this video prior to beginning their colonoscopy preparation. Information to access the YouTube video will be provided to the patients by endoscopy nurse assessment staff when contacting the patients as per standard practice to review appointment scheduling and procedure-day logistics. Group 2 will consist of 30 subjects who will not receive instructions to view the video.

Nursing staff will be asked to grade bowel preps according to the Boston Bowel Preparation Scale (BBPS), a validated and reliable instrument for assessing quality of bowel preparation [6]. Using the BBPS, a four point scoring system is applied to each of the three broad regions of the colon: the right side of the colon (including the cecum and ascending colon), the transverse section of the colon (including the hepatic and splenic flexures), and the left side of the colon (including the descending colon, sigmoid colon, and rectum). The points are assigned as follows: (0), unprepared colon segment, (1), portion of the mucosa of the colon segment seen, (2), minor amount of residual staining, (3), entire mucosa of colon segment seen well. The three segment scores are then summed for a total BBPS score, which ranges from 0 to 9. The maximum BBPS score for a perfectly clean colon without any residual liquid is 9, and the minimum BBPS score for an unprepared colon is 0. The endoscopy nurse who is in the procedure room will be scoring the bowel preparation. This protocol has been employed previously in the VUMC Endoscopy Lab and the endoscopy nurses at Vanderbilt have completed a detailed in-service training session on using the BBPS scoring system. Prior to initiation of this current study protocol, the endoscopy nurses will have a BBPS scoring system review session to ensure continued reliable and valid BBPS scores. The endoscopy nurses will be blinded to whether the patient viewed the video or not.

ELIGIBILITY:
Inclusion Criteria:

* Elective outpatient procedures performed for diagnostic purposes:

  * screening colonoscopy
  * surveillance colonoscopy

Exclusion Criteria:

* Colonoscopy for diagnosis/therapy of acute gastrointestinal hemorrhage or for planned therapeutic intervention
* Colonoscopy performed on hospital inpatients

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation as defined by the Boston Bowel Preparation Scale (total score ≥6 with no score less than 2) | At time of colonoscopy

SECONDARY OUTCOMES:
Bowel preparation quality as defined by the Boston Bowel Preparation Scale (total and segment scores) | At time of colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Keith Obstein, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided